CLINICAL TRIAL: NCT07351825
Title: Prognostic Value of Multiparametric Cardiovascular Magnetic Resonance in Patients With Ischemic Heart Disease: A Multicenter Retrospective Cohort Study
Brief Title: CMR Prognostic Markers in Ischemic Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Beijing Natural Science Foundation (Other)
Responsible Party: Principal Investigator, Minjie Lu, Professor and Director, Department of Cardiovascular Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-IHD; 82471973 (Other Grant/Funding Number: National Natural Science Foundation of China); 7242110 (Other Grant/Funding Number: Beijing Natural Science Foundation); 2022-GSP-QZ-5 (Other Grant/Funding Number: National High Level Hospital Clinical Research Funding)
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Heart Disease (IHD); Myocardial Infarction (MI)
Keywords: Ischemic heart disease; Cardiovascular magnetic resonance; Late gadolinium enhancement; Radiomics; Risk stratification; Prognosis
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic Heart Disease Cohort: Adult patients with ischemic heart disease who underwent clinically indicated cardiac magnetic resonance imaging. Imaging, clinical, and follow-up data are collected for observational analyses, including quantitative imaging, outcome assessment, and exploratory modeling.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Cardiac magnetic resonance imaging performed as part of routine clinical care. Imaging data are used for observational research analyses only, without altering clinical management.

SUMMARY:
Ischemic heart disease (IHD) remains a leading cause of morbidity and mortality worldwide. Accurate risk stratification is essential for guiding clinical management and improving long-term outcomes in patients with ischemic myocardial injury.

Cardiovascular magnetic resonance (CMR) imaging provides comprehensive assessment of myocardial structure, function, and tissue characteristics, enabling detailed evaluation of ischemic injury and its consequences.

This multicenter, retrospective observational study aims to investigate the prognostic value of multiparametric CMR-derived imaging markers in patients with ischemic heart disease who underwent clinically indicated CMR examinations. Imaging parameters of interest include late gadolinium enhancement (LGE), infarct size, microvascular obstruction (MVO), left ventricular and left atrial strain, and native T1 and T2 mapping values.

Long-term clinical outcomes will be obtained from existing medical records. The primary outcome is major adverse cardiovascular and cerebrovascular events (MACCE), and secondary outcome is cardiovascular death. This study seeks to clarify the role of CMR in long-term risk stratification of patients with ischemic heart disease.

DETAILED DESCRIPTION:
This is a multicenter, retrospective observational cohort study based on existing clinical and cardiovascular magnetic resonance (CMR) imaging data. Patients with ischemic heart disease who underwent clinically indicated CMR examinations will be included. Data are derived from multiple centers and span an extended time period, reflecting real-world clinical practice.

CMR examinations were performed as part of routine clinical care. Imaging parameters to be analyzed include late gadolinium enhancement (LGE) for assessment of myocardial scar and ischemic injury, infarct size, presence of microvascular obstruction (MVO), left ventricular and left atrial strain parameters, and native T1 and T2 mapping values when available. Image analysis will be conducted using standardized post-processing methods.

Demographic characteristics, cardiovascular risk factors, treatment strategies, and follow-up data will be collected retrospectively from institutional databases and medical records. The primary outcome of interest is major adverse cardiovascular and cerebrovascular events (MACCE), defined as a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, and unplanned coronary revascularization. The secondary outcome is cardiovascular death.

The primary objective of this study is to evaluate the association between multiparametric CMR-derived imaging markers and long-term clinical outcomes in patients with ischemic heart disease. Secondary objectives include exploring the incremental prognostic value of CMR parameters beyond conventional clinical risk factors and assessing their role in improving individualized risk stratification.

Advanced image analysis techniques, including radiomics and machine learning-based methods, may be applied to CMR images to explore imaging-derived features associated with long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age).
2. Patients with ischemic heart disease, including prior or recent myocardial infarction, who underwent clinically indicated cardiac magnetic resonance (CMR) imaging.
3. Availability of analyzable CMR images, including but not limited to cine imaging, late gadolinium enhancement (LGE), and parametric mapping sequences (T1 and/or T2 mapping), as applicable.
4. Availability of baseline clinical data and longitudinal follow-up information.

Exclusion Criteria:

1. Poor image quality or incomplete CMR data precluding quantitative analysis.
2. Presence of other severe comorbid conditions expected to significantly affect survival or clinical outcomes.
3. Missing key clinical outcome data during follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational study includes adult patients with ischemic heart disease who underwent clinically indicated cardiac magnetic resonance imaging as part of routine clinical care at participating centers. The study population represents a real-world cohort with a broad spectrum of ischemic heart disease, including myocardial infarction, and is characterized by comprehensive CMR imaging data, detailed clinical information, and long-term follow-up for cardiovascular outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events | From the date of index clinically indicated cardiac magnetic resonance imaging to the date of first occurrence of a MACCE event, death, or last available clinical follow-up, whichever came first, assessed up to 10 years.
  Major adverse cardiovascular and cerebrovascular events (MACCE), defined as a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, and unplanned coronary revascularization. Events are identified through longitudinal clinical follow-up and review of medical records.

SECONDARY OUTCOMES:
Cardiovascular Death | From the date of index clinically indicated cardiac magnetic resonance imaging to the date of cardiovascular death or last available clinical follow-up, whichever came first, assessed up to 10 years.
  Death resulting from cardiovascular causes, including myocardial infarction, heart failure, fatal arrhythmia, or sudden cardiac death, as determined by clinical records and follow-up data.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including imaging-derived parameters and relevant clinical variables, will be available upon reasonable request. Data sharing will be considered after publication of the primary results and will require approval by the study investigators and the institutional ethics committee, with a data use agreement in place.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting documents will be available beginning 6 months after publication of the primary results and will remain available for a minimum of 5 years. Access will be granted upon reasonable request, subject to approval by the study investigators and the institutional ethics committee, and execution of a data use agreement.
Access Criteria: Access to individual participant data (IPD) and supporting documents will be granted to qualified researchers with a legitimate scientific proposal. Requests will be reviewed by the study investigators and subject to approval by the institutional ethics committee. Approved users will be required to sign a data use agreement. Data will be shared in a de-identified format via secure data transfer methods. Proposals should be submitted by email to the corresponding investigator.